CLINICAL TRIAL: NCT03272542
Title: Prebiotic Intervention to Improve Calcium Absorption After Gastric Bypass Surgery
Brief Title: PRebiotic to IMprovE Calcium Absorption
Acronym: PRIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anne Schafer, Assistant Professor of Medicine and of Epidemiology and Biostatistics; Staff Physician, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17-22618; R21DK112126 (NIH)
Record Dates: First submitted 2017-08-25; First posted 2017-09-05 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: gastric bypass; calcium absorption; postmenopausal women
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled pilot trial with a parallel-arm design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic: soluble corn fiber (Experimental): SCF (PromotorTM Soluble Corn Fiber 85, provided by manufacturer Tate & Lyle) will be dispensed to participants as a dry powder in sachets of 12 g SCF85 product (which is approximately 10 g fiber). Participants will mix the powder into 250 mL water and consume two such beverages daily, ≥1 hour apart. (For the first week, all participants will consume one beverage daily, and subsequently increase to one beverage twice daily.) Participants will be asked to substitute these for 500 mL of their usual daily water intake but to make no other dietary changes.
  Interventions: Dietary Supplement: Prebiotic: soluble corn fiber
- Placebo (Placebo Comparator): The placebo control will be maltodextrin powder in identical sachets. Participants will mix the powder into 250 mL water and consume two such beverages daily, ≥1 hour apart. (For the first week, all participants will consume one beverage daily, and subsequently increase to one beverage twice daily.) Participants will be requested to substitute these for 500 mL of their usual daily water intake but to make no other dietary changes.
  Interventions: Dietary Supplement: Placebo: maltodextrin

INTERVENTIONS:
Dietary Supplement: Prebiotic: soluble corn fiber — prebiotic
  Other Names: PROMOTOR 85
  Arms: Prebiotic: soluble corn fiber
Dietary Supplement: Placebo: maltodextrin — placebo
  Arms: Placebo

SUMMARY:
Gastric bypass surgery is a highly effective treatment for obesity, but it has negative effects on skeletal health, due in part to a dramatic decline in intestinal calcium absorption capacity. Animal and human studies suggest that non-digestible fibers termed prebiotics, such as soluble corn fiber (SCF), augment calcium absorption in the lower intestine as they act as substrates for beneficial gut microbiota. This is a pilot randomized controlled trial of the effects of SCF vs. placebo on intestinal calcium absorption, bone turnover marker levels, and the gut microbiome in postmenopausal women who have previously undergone gastric bypass surgery.

DETAILED DESCRIPTION:
The study is a pilot randomized control trial (RCT) of the effects of the prebiotic SCF vs. placebo in 20 postmenopausal women who underwent Roux-en-Y gastric bypass surgery 2-6 years previously and thus have completed the postoperative period of rapid weight loss and metabolic and dietary change. A 24 g/day dose of SCF85 (which is approximately 20 g/day fiber) will be tested, as that dose was proven effective for calcium absorption/retention in healthy postmenopausal women and adolescents. The SCF and the maltodextrin placebo will be mixed in water and consumed in divided doses twice daily for 2 months, a duration exceeding other SCF trials but remaining feasible for a pilot. The primary outcome will be change in intestinal calcium absorption, which is the efficacy outcome about which the study must collect preliminary data and from which the investigators must refine power calculations for the anticipated future trial. Because the investigators hypothesize that an increase in calcium absorption will decrease bone turnover and ultimately increase bone mineral density (BMD), the study will measure biochemical markers of bone turnover in this pilot. Secondary outcomes will be gastrointestinal tolerability and acceptability. On an exploratory basis, the study will determine effects of the prebiotic on the gut microbiome. This pilot will yield critical experience about feasibility of recruitment and adherence to the intervention and measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women (no menses for ≥4 yrs)
2. ≤ 75 yrs old,
3. Underwent Roux-en-Y gastric bypass surgery for weight loss 2-6 years prior

Exclusion Criteria:

1. Serum 25(OH)vitamin D level <30 ng/mL (to remove the effect of vitamin D insufficiency/deficiency)*
2. History of >1 bariatric surgical procedure
3. Antibiotic therapy in the last 3 months
4. Regular pre- or probiotic use in the last 3 months
5. Regain of >50% of weight loss post-bypass
6. Calculated creatinine clearance <30 mL/min
7. Serum calcium >10.2 mg/dL
8. Use of hormone therapy, osteoporosis pharmacotherapy, glucocorticoids, or other medications impacting calcium metabolism
9. Thyroid stimulating hormone (TSH) <0.01 milli-international units per liter (mIU/L)

A potential participant may be excluded if she has a condition or abnormality that in the opinion of the Investigator would compromise the safety of the participant or the quality of the data.

*Women excluded due to 25(OH)D level will be offered re-screening after vitamin D supplementation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in fractional intestinal calcium absorption | 2 months
  Fractional calcium absorption to be determined using dual stable isotopic tracers

SECONDARY OUTCOMES:
Change in bone turnover markers | 2 months
  Serum biochemical markers of bone turnover C-telopeptide (CTX) and procollagen type 1 N-terminal propeptide (P1NP)
Gastrointestinal tolerability | 2 months
  Self-reported flatulence, bloating, abdominal pain, stomach noises
Acceptability | 2 months
  Self-reported satisfaction, likelihood that one would be willing to consume the beverage for 12 months
Change in gut microbiome composition | 2 months
  Stool bacterial and fungal composition to be analyzed, including alpha diversity and beta diversity metrics as well as taxon relative abundance, with subsequent in silico metagenomic predictions of enrichment of bacterial functional gene pathways

CONTACTS AND LOCATIONS:
Overall Officials: Anne Schafer, MD, Principal Investigator — UCSF & SFVAMC
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu KC, Cao S, Weaver CM, King NJ, Patel S, Kingman H, Sellmeyer DE, McCauley K, Li D, Lynch SV, Kim TY, Black DM, Shafer MM, Ozcam M, Lin DL, Rogers SJ, Stewart L, Carter JT, Posselt AM, Schafer AL. Prebiotic to Improve Calcium Absorption in Postmenopausal Women After Gastric Bypass: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2022 Mar 24;107(4):1053-1064. doi: 10.1210/clinem/dgab883. PMID 34888663